CLINICAL TRIAL: NCT01634022
Title: Effectiveness of Acupuncture on Treating Major Depressive Disorder
Brief Title: Effectiveness of Acupuncture for Depressed Patients Not Taking Antidepressant Medications
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Albert Yeung, Director of Primary Care Research, Depression Clinical and Research Program, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2004P002819
Record Dates: First submitted 2012-06-15; First posted 2012-07-06 (Estimated); Last update posted 2012-07-06 (Estimated); Status verified 2012-07

CONDITIONS: Depression
Keywords: Acupuncture; Antidepressant; Monotherapy; Depression; Alternative treatments
MeSH Terms: conditions — Depression | interventions — Acupuncture Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Acupuncture (Experimental): Adults with depression who are not currently taking an antidepressant medication.
  Interventions: Procedure: Acupuncture

INTERVENTIONS:
Procedure: Acupuncture — 5 specific body acupoints (HT-7 and LI-4 on the hands bilaterally, and ST-36, SP-6, and LR-3 on the legs bilaterally) with gentle manual tonification every 10 min. Two acupoints along the midline of the head, GV-20 and GV-24.5 (Yintang), were also used with a 2 Hz current applied from GV-20 (-) to GV24.5 (+).

SUMMARY:
Acupuncture is a popular complementary/alternative therapy that has been in use for thousands of years for the treatment of various medical and psychiatric conditions, including Major Depressive Disorder (MDD). In this study, the investigators applied the investigators acupuncture-treatment-for-depression protocol, based on Traditional Chinese Medicine (TCM) principles for treating MDD, to depressed patients not taking any antidepressant medications (a protocol that the investigators previously piloted as a medication augmentation therapy for partial responders with MDD).

The investigators specifically investigated the efficacy, safety, and tolerability of this TCM-based protocol for such patients, as well as potential differences in outcomes between weekly vs. twice-weekly treatment. The investigators hypothesized that acupuncture monotherapy would be associated with a response rate of at least 50%, which the investigators defined as a decrease in depressive symptoms from the beginning to the end of the study of 50% or more, and that the response would be greater among patients who received acupuncture 2 times per week (vs. 1 time per week). The investigators also hypothesized that acupuncture would be associated with minimal side effects.

ELIGIBILITY:
Inclusion Criteria:

* Has current or past DSM-IV MDD diagnosis based on SCID; AND current 17-Hamilton Rating Scale for Depression (BRSD) score of 14 or above
* Age between 18-65
* No treatment with antidepressant(s) in the past 3 months
* If patient has received psychotherapy, no initiation or termination of therapy in the past 3 months.

Exclusion Criteria:

* Patients with primary diagnosis other than Major Depressive Disorder, or any history of psychosis or mania.
* Conditions that could make it difficult to conclusively determine that depressive symptoms were the result of MDD and not some other condition, including substance abuse or dependence within the last 6 months, medical conditions that could produce depression, including epilepsy, history of an abnormal EEG, severe head trauma, or stroke.
* Serious uncontrolled medical conditions [e.g. poorly controlled diabetes, severe congestive heart failure], or other medical conditions that have not been stable for at least 3 months.
* Electroconvulsive therapy (ECT) during the last year.
* Current active suicidal or self-injurious potential necessitating immediate treatment.
* Currently receiving concomitant Acupuncture Treatment, or any Acupuncture treatment in the past three months.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2005-05; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Change in scores on the Hamilton Depression Rating Scale, 17 items (HAM-D-17) | Baseline and all acupuncture sessions (weekly) for 8 weeks
  The HAM-D-17 is a clinician-rated assessment (structured interview) of patients' depressive symptoms. Questions focus on depressive symptoms during the past 7 days, and higher cumulative scores (possible responses to each item range from 0-4 or 0-2) indicate more severe depression.

SECONDARY OUTCOMES:
Response to treatment, defined as a 50% or greater improvement in HAM-D-17 score compared to baseline | Baseline and all acupuncture sessions (weekly) for 8 weeks
  (See primary outcome measure description.)

CONTACTS AND LOCATIONS:
Overall Officials: Albert Yeung, MD, ScD, Principal Investigator — Depression Clinical and Research Program, Massachusetts General Hospital
Locations (1):
- Depression Clinical and Research Program, Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Result] Mischoulon D, Brill CD, Ameral VE, Fava M, Yeung AS. A pilot study of acupuncture monotherapy in patients with major depressive disorder. J Affect Disord. 2012 Dec 10;141(2-3):469-73. doi: 10.1016/j.jad.2012.03.023. Epub 2012 Apr 21. PMID 22521855